CLINICAL TRIAL: NCT06551636
Title: Effects on the Expiratoriy Flow of Assisted Autogen Drainage in a Critical Patient Wtih Invasive Mechanical Ventilation
Brief Title: Effects on the Expiratory Flow of AAD in a Critical Patient With IMV
Status: Completed | Type: Observational
Sponsor: Parc Taulí Hospital Universitari (Other)
Responsible Party: Principal Investigator, julia estela, Msc PT, Parc Taulí Hospital Universitari
Other Study IDs: 2019685
Record Dates: First submitted 2024-05-20; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Respiratory Physiotherapy
Keywords: respiratory physiotherapy; invasive ventilation; critical care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: respiratory physiotherapy (AAD) — The AAD technique involves placing the physiotherapist's hands on the chest where the secretions are identified and applying pressure to the chest. The maneuver will last according to the patient's tolerance, in an average of approximately 10 min.

SUMMARY:
One of the detrimental effects of invasive mechanical ventilation (IMV) is the alteration of the patient's mucociliary system that requires ventilatory support. The consequence of poor drainage of secretions, triggers secretion retention, atelectasis, and ventilator-associated pneumonia (VAP). Respiratory physiotherapy in the intubated patient facilitates the mobilization of retained and impacted secretions in the bronchial tree, decreasing resistance, improving lung compliance, and decreasing respiratory muscle work.

The main objective of the present study is to measure the expiratory flow generated by the application of the DAA technique in the intubated patient during, after, at the end of the technique and at two hours. As secondary objectives, it is proposed to observe whether the application of the DAA maneuver in the patient with IMV improves oxygenation, produces changes in respiratory mechanics, improves air entrapment, decreases exhaled volume post DAA and analyzes the tolerance of DAA in IMV-conscious patients The study will be performed on patients admitted to the Intensive Care Unit (ICU) of the Parc Taulí University Hospital in Sabadell with IMV requirements. The intervention will consist of performing a respiratory physiotherapy session as usual in the daily clinical practice of the ICU, specifically the technique of assisted autogenous drainage, before, during and after the Better CareTM platform will be used to continuously record the physiological variables. necessary for the study.

DETAILED DESCRIPTION:
Ventilated air blown into the bronchial shaft through the orotracheal tube (OT) causes ciliary dyskinesia by decreasing the rate of progression of secretions to the proximal pathways. The consequence of poor drainage of secretions is triggered by retention of secretions, atelectasis, and ventilator-associated pneumonia (VAP).

Humidification and heating of the air with devices added to the imv together with respiratory physiotherapy aim to prevent and / or treat respiratory complications. Respiratory physiotherapy in the intubated patient facilitates the mobilization of retained and impacted secretions in the bronchial tree, helping to decrease resistance, improve lung compliance, and decrease respiratory muscle work.

Respiratory physiotherapy consists of a variety of devices and manual techniques to improve secretion drainage, ventilatory mechanics, and gas exchange.

The lack of scientific evidence on the effect and efficacy of respiratory physiotherapy in the patient with imv makes it difficult for the physiotherapist to perform his task with certainty of the impact of the intervention on lung physiology. Published clinical guidelines recommend the application of respiratory physiotherapy techniques to critically ill patients, but the need to demonstrate their effects with well-designed, quality studies and conclusive results is emphasized.

The aim of this study is to analyze the effect of the technique developed by the Belgian physiotherapist Jean Chevaillier, called assisted autogen drainage (AAD), on the intubated patient.

AAD is defined as a secretion drainage technique where the goal is to create a sufficiently sustained, homogeneous and synchronous expiratory flow, increasing speed, and seeking an erosion effect on secretions at different levels of the bronchial tree.

In the review of the literature on respiratory physiotherapy in the area of critics and in patients with IMV, articles have been found with different techniques such as hyperinsufflation, techniques for increasing the expiratory flow such as squeezing or rib cage. compression ". These demonstrate the safety of the techniques but there is controversy over the effect of maneuvers on the drainage of secretions and ventilatory mechanics. The point of discussion in the discussion of the authors of the meta-analyzes and studies is the need for new studies evaluating the effectiveness of respiratory physiotherapy in lung mechanics.

Hypothesis Respiratory physiotherapy applied through assisted autogenous drainage increases respiratory flow in the airways and therefore may modify respiratory mechanics and promote drainage in ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

* The subjects will be all patients over the age of 18 who are admitted to the ICU of the Parc Taulí University Hospital in Sabadell with IMV requirements
* Subjects with hemodynamic stability; Higher mean blood pressure (PAM) 65 mmg, Heart rate (HR) less than 110 bpm and Oxygen saturation (SpO2) greater than 90% with or without norepinephrine <0.5 mcg / Kg / min.

Exclusion Criteria:

* patients with platelet pressures (Pm) greater than 30 cmH2O and / or expiratory pressure at the end of expiration (PEEP) ≥ 10cmH2O
* patients who carriers of thoracic drainage
* patients with costal and / or sternal fractures
* pneumothorax
* pregnant women
* Obesity (BMI> 35)
* agitated patients with RASS greater than or equal to 3
* patients with intracranial pressures greater than 20 cmH2O
* dying.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The subjects will be all patients over the age of 18 who are admitted to the ICU of the Parc Taulí University Hospital in Sabadell with IMV requirements
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
To measure the expiratory flow in the intubated patient | Data will be collected, 10 minutes (one hour before intervention), during 10 minutes (time of the respiratory physiotherapy session) and 10 min, two hours after therapy.
  The following physiological variables will be obtained through the BC Link software using the services of the I3PT signal laboratory: final expiratory flow 25-75%(L/min)

SECONDARY OUTCOMES:
To observe if the application of the AAD maneuver improves, produces changes in the respiratory mechanics; Compliance; Cst= Vt/Pplat-PEEP (ml/cmH2O) | Data will be collected, 10 minutes (one hour before intervention), during 10 minutes (time of the respiratory physiotherapy session) and 10 min, two hours after therapy.
  The following physiological variables will be obtained through the BC Link software, re using the services of the I3PT signal laboratory.
To observe if the application of the AAD maneuver improves, produces changes in the respiratory mechanics; Resistance R=Ppeak-Pplat/flow ( kPa x L-1 x sg) | Data will be collected, 10 minutes (one hour before intervention), during 10 minutes (time of the respiratory physiotherapy session) and 10 min, two hours after therapy.
  The following physiological variables will be obtained through the BC Link software, re using the services of the I3PT signal laboratory.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Parc Taulí, Sabadell, Barcelona, Spain

REFERENCES:
- [Background] Konrad F, Schreiber T, Brecht-Kraus D, Georgieff M. Mucociliary transport in ICU patients. Chest. 1994 Jan;105(1):237-41. doi: 10.1378/chest.105.1.237. PMID 8275739
- [Background] Pneumatikos IA, Dragoumanis CK, Bouros DE. Ventilator-associated pneumonia or endotracheal tube-associated pneumonia? An approach to the pathogenesis and preventive strategies emphasizing the importance of endotracheal tube. Anesthesiology. 2009 Mar;110(3):673-80. doi: 10.1097/ALN.0b013e31819868e0. PMID 19212256
- [Background] Pattanshetty RB, Gaude GS. Effect of multimodality chest physiotherapy on the rate of recovery and prevention of complications in patients with mechanical ventilation: a prospective study in medical and surgical intensive care units. Indian J Med Sci. 2011 May;65(5):175-85. PMID 23364504
- [Background] Spapen HD, De Regt J, Honore PM. Chest physiotherapy in mechanically ventilated patients without pneumonia-a narrative review. J Thorac Dis. 2017 Jan;9(1):E44-E49. doi: 10.21037/jtd.2017.01.32. PMID 28203436
- [Background] Branson RD. Secretion management in the mechanically ventilated patient. Respir Care. 2007 Oct;52(10):1328-42; discussion 1342-7. PMID 17894902
- [Background] Volsko TA. Airway clearance therapy: finding the evidence. Respir Care. 2013 Oct;58(10):1669-78. doi: 10.4187/respcare.02590. PMID 24064626
- [Background] Ambrosino N, Janah N, Vagheggini G. Physiotherapy in critically ill patients. Rev Port Pneumol. 2011 Nov-Dec;17(6):283-8. doi: 10.1016/j.rppneu.2011.06.004. Epub 2011 Jul 22. PMID 21782380
- [Background] Calvo-Ayala E, Khan BA, Farber MO, Ely EW, Boustani MA. Interventions to improve the physical function of ICU survivors: a systematic review. Chest. 2013 Nov;144(5):1469-1480. doi: 10.1378/chest.13-0779. PMID 23949645
- [Background] Guimaraes FS, Lopes AJ, Constantino SS, Lima JC, Canuto P, de Menezes SL. Expiratory rib cage Compression in mechanically ventilated subjects: a randomized crossover trial [corrected]. Respir Care. 2014 May;59(5):678-85. doi: 10.4187/respcare.02587. Epub 2013 Oct 8. PMID 24106324
- [Background] Borges LF, Saraiva MS, Saraiva MAS, Macagnan FE, Kessler A. Expiratory rib cage compression in mechanically ventilated adults: systematic review with meta-analysis. Rev Bras Ter Intensiva. 2017 Jan-Mar;29(1):96-104. doi: 10.5935/0103-507X.20170014. PMID 28444078
- [Background] Gosselink R, Bott J, Johnson M, Dean E, Nava S, Norrenberg M, Schonhofer B, Stiller K, van de Leur H, Vincent JL. Physiotherapy for adult patients with critical illness: recommendations of the European Respiratory Society and European Society of Intensive Care Medicine Task Force on Physiotherapy for Critically Ill Patients. Intensive Care Med. 2008 Jul;34(7):1188-99. doi: 10.1007/s00134-008-1026-7. Epub 2008 Feb 19. PMID 18283429